CLINICAL TRIAL: NCT01394718
Title: Analgesia Efficacy of Repeated Doses of Intravenous Acetaminophen (Paracetamol) in the Pediatric Spinal Fusion Population
Brief Title: Analgesic Efficacy of Repeated Doses of Intravenous (IV) Acetaminophen in Post-operative Pediatric Spine Fusion Patients
Acronym: IV APAP SF
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Children's Hospital of Philadelphia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 11-08095
Record Dates: First submitted 2011-07-13; First posted 2011-07-14 (Estimated); Results first posted 2016-04-18 (Estimated); Last update posted 2016-04-18 (Estimated); Status verified 2016-03

CONDITIONS: Pain, Postoperative
Keywords: analgesic adjunct; acetaminophen; spine fusion surgery; opiate reduction; pain management after elective surgical operation
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Saline Placebo (Placebo Comparator): Control subjects will receive saline as placebo at the time of skin closure intra-operatively and will continue to receive IV saline for 44 hours post-operatively. Doses will be administered every 6 hours (total of 8 doses).
  Interventions: Other: Placebo
- Intravenous Acetaminophen (Experimental): Subjects will receive the first dose of intravenous (IV) acetaminophen (at 15 mg/kg, with maximum doses based on patient age and weight) at the time of skin closure intra-operatively and will continue to receive IV acetaminophen for 42 hours post-operatively. Doses will be administered every 6 hours (total of 8 doses).
  Interventions: Drug: Intravenous Acetaminophen

INTERVENTIONS:
Drug: Intravenous Acetaminophen — Scheduled doses of 15 mg/kg of IV acetaminophen will be administered to the treatment arm of the study for a total of 8 doses over a 48 hour period post-operatively.
  Arms: Intravenous Acetaminophen
Other: Placebo — Saline placebo will be given at the time of skin closure intra-operatively and will continue to receive IV saline for 44 hours post-operatively. Doses will be administered every 6 hours (total of 8 doses).
  Arms: Saline Placebo

SUMMARY:
This is a prospective, randomized, double-blinded, placebo controlled trial Potential subjects will be identified from the Pre-Surgical Anesthesia Clinic visit. Parents/legal guardians will be approached about study participation at the Anesthesia outpatient pre-visit. Attending Anesthesiologist will receive e-mail notification about potential subject participation the day before the scheduled surgery. Study lab (hepatic function panel) will be collected as soon as possible after anesthesia induction by anesthesia. Results will be reviewed by study team member and study drug will be ordered by study team if patient does not meet exclusion criteria. Study drug (IV acetaminophen or placebo) will be administered at the time of skin closure by anesthesia on completion of the surgical procedure (after randomization). Study drug will be administered every 6 hours for 2 days. Subjects will continue to receive standard of care with patient controlled analgesia (PCA) opiate therapy (morphine or hydromorphone) for analgesia as per the Pain Management Service. Pain scores, opiate (morphine equivalent) administered, requirements for treatment of opiate related side effects (treatment for nausea and itching), and certain post-operative characteristics will be measured for up to 4 days post-operatively (time to mobilization, time to diet advancement, time to discharge).

DETAILED DESCRIPTION:
An ideal drug as an opiate-sparing analgesic adjunct, acetaminophen, unlike some other drugs, is platelet function sparing, and thus particularly useful in the post-operative orthopedic patient population. In part because of its well established safety profile, as well as minimal drug interactions, acetaminophen is considered a cornerstone of a multimodal analgesic approach. Several studies have described the clinically significant beneficial effects of a multimodal drug approach to analgesia, citing improved pain control and a shorter recovery time. Reduced adverse events and improved pain control with multimodal analgesia drug approaches may result in shorter hospitalizations, improved recovery and function, and reduced health care costs. Opiate therapy, while effective analgesia, is associated with a variety of potential adverse side effects, including pruritus, nausea, emesis, ileus, respiratory depression, tolerance, addiction and sedation. These adverse effects may limit post-operative mobility, postpone return of bowel function, cause feeding intolerance, prolong hospitalization, and postpone post-operative recovery.

While oral acetaminophen is useful as an opiate-sparing therapy, the oral route of drug administration may not be feasible in the early post-operative period. Enteral drug absorption in the initial post-operative period may be erratic, with negative impacts on therapeutic effect. Intravenous acetaminophen may a particularly useful analgesic in these circumstances. At present, there are no pediatric studies in the United States examining the efficacy of multiple- dose IV acetaminophen in the post-operative surgical population. This study will compare analgesic efficacy, nausea and pruritus scores, time to recovery, and length of hospital stay in two subject groups who are status post spine fusion surgery: those who receive schedule IV acetaminophen and opiate for 48 hours, and those who are treated with standard opiate therapy without IV acetaminophen.

ELIGIBILITY:
Inclusion Criteria:

Subjects 10-18 years who are status post anterior or posterior spine fusion surgery

Exclusion Criteria:

1. All patients requiring mechanical ventilation post-operatively, continuous infusions of sedative, or continuous infusions of alternate opiates (i.e. fentanyl)
2. Patients with hepatic dysfunction
3. Patients with chronic opiate requirements
4. Pregnant or lactating females
5. Patients placed on opiates other than morphine or hydromorphone
6. Patients with opiate or acetaminophen allergies
7. Patients placed on alternate analgesic adjuncts (i.e. ketamine, etc)
8. Patients who receive intrathecal opiates

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 67 (Actual)
Dates: Start 2011-07; Primary Completion 2014-06 (Actual); Study Completion 2015-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Athena Zuppa, MD, Principal Investigator — Children's Hospital of Philadelphia
Locations (1):
- Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All children of ages 10-18 undergoing posterior spine fusion surgery for idiopathic or neuromuscular scoliosis between July 2011 and May 2014 were eligible for inclusion.
Pre-assignment Details: 281 subjects were screened, 125 approached for consent/assent and 67 consented/assented. Of the initial 67 subjects, 1 was withdrawn by the clinical team, 1 patient's surgery was cancelled, 2 were withdrawn by the family, and 3 were deemed ineligible after consent were removed from the study.
Period: Overall Study
Arm/Group | Saline Placebo | Intravenous Acetaminophen
Started | 30 | 30
Completed | 28 | 29
Not Completed | 2 | 1
Not completed — Met protocol-specific stopping criteria | 2 | 1

BASELINE CHARACTERISTICS:
Population: Analysis population includes only those subjects who completed at least 24 hours of post-operative data collection. 3 subjects who were enrolled and received at least 1 dose were removed before reaching the 24 hour post-operative milestone.
Groups:
- Total: Total of all reporting groups
Arm/Group | Saline Placebo | Intravenous Acetaminophen | Total
Number analyzed (Participants) | 28 | 29 | 57
Age, Continuous [Mean (Standard Deviation); unit: years] | 14.43 (1.69) | 14.17 (1.87) | 14.30 (1.77)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 25 | 44
  Male | 9 | 4 | 13
Region of Enrollment [Number; unit: participants]
  United States | 28 | 29 | 57
Weight [Mean (Standard Deviation); unit: kilograms (kg)] | 59.79 (13.69) | 53.44 (11.32) | 56.56 (12.83)
Surgery Duration [Mean (Standard Deviation); unit: hours (hr)] | 5.21 (1.03) | 5.09 (1.14) | 5.15 (1.08)
Estimated Blood Loss (EBL) [Median (Full Range); unit: milliliter (ml)] | 775 [450 to 2200] | 600 [150 to 1400] | 700 [150 to 2200]
Intra-operative methadone [Median (Full Range); unit: milligrams (mg)] | 6.3 [0 to 10] | 6.0 [0 to 10] | 6.0 [0 to 10]
Intra-operative methadone [Median (Full Range); unit: milligrams/kilograms (mg/kg)] | 0.1 [0 to 0.2] | 0.1 [0 to 0.2] | 0.1 [0 to 0.2]

OUTCOME MEASURES:

1. Primary Outcome: Total Opiate Requirement
Description: Total opiate requirement was monitored 24 hours post-operatively. Morphine and hydromorphone measurements were totaled and recorded in mg/kg/day of morphine equivalents.
Time Frame: 24 hours
Population: Subjects were deemed evaluable if a minimum of 24 hours of data was collected post-operatively, with receipt of at least four doses of study drug, prior to study withdrawal or unblinding, with T0 (time zero) being time of administration of first dose of either treatment drug or placebo.
Measure: Mean (Standard Deviation); unit: mg/kg
Arm/Group | Saline Placebo | Intravenous Acetaminophen
Number analyzed (Participants) | 28 | 29
mg/kg | 1.19 (0.43) | 1.01 (0.32)

2. Secondary Outcome: Average Pain Score
Description: Pain Scores were monitored using the numeric pain assessment scale in both treatment arms of the study and recorded and averaged for the first 24 hours after initial intra-operative dose of study drug. The numeric pain assessment scale is a verbal self-reported pain assessment that ranges between 1 (no pain) to 10 (worst pain imaginable).
Time Frame: 24 hours
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Saline Placebo | Intravenous Acetaminophen
Number analyzed (Participants) | 28 | 29
units on a scale | 4.53 (2.02) | 4.62 (1.99)

3. Secondary Outcome: Average Nausea Score
Description: Nausea scores were recorded by the nursing staff approximately 4 times over the first 24 hours and then averaged for the 24 hour period. Nausea Scores range from 1 (none) to 4 (severe).
Time Frame: 24 hours
Population: as for outcome 1
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Saline Placebo | Intravenous Acetaminophen
Number analyzed (Participants) | 28 | 29
units on a scale | 1.2 [1.0 to 2.5] | 1.0 [1.0 to 2.6]

4. Secondary Outcome: Average Pruritus Score
Description: Pruritus scores were recorded by the nursing staff approximately 4 times over the first 24 hours and then averaged for the 24 hour period. Pruritus scores range from 1 (none) to 3 (intolerable).
Time Frame: 24 hours
Population: as for outcome 1
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Saline Placebo | Intravenous Acetaminophen
Number analyzed (Participants) | 28 | 29
units on a scale | 1.0 [1.0 to 2.5] | 1 [1.0 to 2.0]

ADVERSE EVENTS:
Time Frame: 96 Hours
Arm/Group | Saline Placebo | Intravenous Acetaminophen
Serious Adverse Events (participants affected / at risk) | 0/28 | 0/29
Other Adverse Events (participants affected / at risk) | 0/28 | 0/29

LIMITATIONS AND CAVEATS:
This is a single center study with subjects confined to a single surgical procedure with a small sample size, possibly limiting generalizability of results.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes